CLINICAL TRIAL: NCT06963697
Title: Expanded Access To Neoantigen Synthetic Long Peptide Vaccines in Patients With Local Or Metastatic Solid Tumors
Status: Available | Type: Expanded Access
Sponsor: Jaime Leandro Foundation for Therapeutic Cancer Vaccines (Other)
Responsible Party: Sponsor
Other Study IDs: JLF-100
Record Dates: First submitted 2023-02-20; First posted 2025-05-09 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Expanded Access Types: Individual, Intermediate

INTERVENTIONS:
Biological: Personalized Synthetic Long Peptide Vaccine — Neoantigen synthetic long peptide vaccines are composed of synthetic long peptides which are 8-35 amino acids in length and designed to induce immune responses to cancer neoantigens identified by exome sequencing. Neoantigen synthetic long peptide vaccines will be co-administered with poly-ICLC, an innate immune adjuvant capable of activating TLR3 and other pathways.

SUMMARY:
This is an intermediate patient expanded access protocol for treatment of patients with local or metastatic solid tumors with a neoantigen synthetic long peptide vaccine.

ELIGIBILITY:
Patients must satisfy the following criteria to be enrolled in the protocol:

Main Inclusion Criterion:

1. Patient who qualifies for treatment under 21 CFR 312.305 based on treating physician judgment, inability to enroll in study JLF-200, must have received or be ineligible for FDA-approved therapies for their specific cancer type, and an estimated 5-year survival of less than 50%.

Other Inclusion Criteria:

1. >= 12 years of age.
2. ECOG performance status ≤ 2 or Karnofsky score of >=70.
3. Adequate organ function allowing favorable benefit to risk ratio per the treating physician
4. Systemic corticosteroid therapy is permitted provided dosing is no greater than 4 mg per day (dexamethasone or equivalent) on the day of vaccine administration.
5. Ability to understand and willingness to sign an IRB approved written informed consent document.

Exclusion Criteria:

1. History of serious adverse reaction to vaccines such as anaphylaxis, hives, or respiratory difficulty or known allergy to a component of the neoantigen synthetic long peptide vaccine.
2. Intercurrent illness requiring chronic use of medications that may interfere with rescue medications for treatment of vaccine-related anaphylaxis or attenuate immune response to vaccine treatment (immunosuppressive therapies).
3. Psychiatric illness or social situations that would limit compliance with study requirements.
4. History of pre-existing immunodeficiency disorder or autoimmune condition requiring immunosuppressive therapy that would preclude response to vaccine. 5. Females of childbearing potential may participate provided they agree to practice abstinence; and, if heterosexually active, agree to use at least 2 highly effective contraceptive methods throughout the study and for 3 months following the last dose of study drug; and have a negative serum pregnancy test.

6. Females of non-childbearing potential must be post-menopausal or have been surgically sterilized.

7. Male subjects with a female partner of childbearing potential must agree to practice abstinence or to use a physician-approved contraceptive method throughout the study and for 3 months following the last dose of study drug.

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Oncology, Austin, Texas, United States